CLINICAL TRIAL: NCT02734589
Title: Fecal Transplantation Using a Novel Conditioning Method for Donor and Recipient in Mild to Moderate Treatment Refractory Colitis in Inflammatory Bowel Disease
Brief Title: Fecal Transplantation Using a Diet for Donor and Recipient in Refractory Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommendation of stopping the trial after reviewing the interim data
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0070-15
Record Dates: First submitted 2016-03-28; First posted 2016-04-12 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Nutrition; microbiome
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fecal microbiota transplantation (FMT) without Diet (Active Comparator): undergo standard fecal transplantation by colonoscopy on day 1 and 60 ml rectal enemas on days 2 and 14 from the same donor without dietary conditioning.
  Interventions: Other: Fecal transplantation
- FMT with Diet for the donor and for the recipient (Experimental): undergo standard fecal transplantation by colonoscopy on day 1 and 60 ml rectal enemas on days 2 and 14 with dietary pre-conditioning of the donor for 14 days and dietary treatment of the recipient immediately after transplantation and for the following 12 weeks.
  Interventions: Other: Unique novel Diet for UC and Unique novel Diet for the donor + FMT
- Dietary therapy only (Active Comparator): The patient will receive detailed instructions regarding the UC diet to be used over 12 weeks without FMT.
  Interventions: Other: Unique novel Diet for UC

INTERVENTIONS:
Other: Fecal transplantation — Transplantation of fecal bacteria from a healthy individual into a recipient- ulcerative colitis patient via colonoscopy and enemas
  Other Names: Fecal microbiota transplantation (FMT)
  Arms: Fecal microbiota transplantation (FMT) without Diet
Other: Unique novel Diet for UC and Unique novel Diet for the donor + FMT — A developed unique diet that is geared to induces remission and decreases inflammation in patients with active UC. Also a conditioning diet for healthy subjects to be used by the donor prior to transplantation- a developed unique diet for two weeks.
  Other Names: Ulcerative Colitis Diet (UCD) and the conditioning diet
  Arms: FMT with Diet for the donor and for the recipient
Other: Unique novel Diet for UC — A developed diet that is geared to induces remission and decreases inflammation in patients with active UC.
  Other Names: Ulcerative Colitis Diet (UCD)
  Arms: Dietary therapy only

SUMMARY:
Changing the microbiota has become the most intriguing target for intervention in inflammatory bowel disease (IBD). Dietary therapy is successful in mild to moderate Crohn's disease and may be effective in mild to moderate ulcerative colitis (UC) as well, though dietary interventions in UC are just getting underway. However these interventions are less likely to be effective for the more severely inflamed or refractory end of the spectrum. Fecal transplantation (FT) has been suggested as a method to treat refractory IBD, but most studies have been unsuccessful in establishing remission and especially sustained remission. The investigators hypothesize that this is due to selection of random donors and the inability to maintain an optimal microbiota eco system post transplant. Diet is a powerful tool to modulate the microbiota. The investigators propose that use of a donor and recipient diet designed for UC during fecal transplantation will be superior to diet alone of fecal transplantation alone and will improve patient outcomes.The investigators propose to modify FT using a novel protocol and approach that we have developed. We have developed a unique diet that is geared to rectify dysbiosis in UC and damage to the mucous layer in active UC. The investigators intend to condition both donor and recipient with the diet to achieve optimal conditions for transplant to succeed for both donor and recipient .The investigators intend to evaluate this protocol in adults with active UC that are refractory to medications. The investigators will start with a randomized controlled trial involving 76 transplanted patients+ 20 subjects for dietary controls with the UC diet alone.

DETAILED DESCRIPTION:
Study type- It will be an open label 3 arm multicenter randomized controlled single blinded study, with review of endoscopic activity by blinded reviewers. Patients will be randomized to one of three groups; Group 1 will undergo standard fecal transplantation by colonoscopy on day 1 and 60 ml rectal enemas on days 2 and 14 from the same donor without dietary conditioning, while Group 2 will undergo the same transplantation (colonoscopy and enemas at night day 2 and day 14), with dietary pre-conditioning of the donor for 14 days and dietary treatment of the recipient immediately after transplantation and for the following 12 weeks.We will attempt to use the same donors for group 1 and 2 by using the preconditioning stool for group 1 and the post conditioning stool for group 2 in order to control for the "donor effect". Group 3 will receive dietary therapy only.Physicians will be blinded to treatment arm and donors used within the transplantation arms. A data safety monitoring board will review safety after the first 34 patients to make sure that there is no ethical problem with continuing the study. The investigators will continue the fecal transplantation trial to reach our target enrolment number ( 76 patients) for transplantation + 20 dietary controls.

Subjects may continue their stable medications but should not start new medications during the 8 week period unless they fail to respond. Steroid weaning can commenced from day 14.

Patients will be seen on weeks0, 2, 6, 8, 12 and during week 20. Week 6 will be only a dietitian visit. The last visit is a visit off diet to evaluate sustainability of the initial intervention, safety and changes in BMI due to FT or diet. A telephone conversation to assess SCCAI will be made at week 1 and week 7. At each visit (weeks 0, 2, 6, 8, 12, 20) patients will have Weight, a disease activity score, PGA, CBC, CRP, albumin and complete chemistry panel performed. Adverse events and medications used will be recorded at each visit.Stool samples for microbiome (16S rDNA, Short chain fatty acid analysis) and Calprotectin will be measured locally at baseline, weeks 2, 8 and 12. All patients (patients in group 1,2 and 3) will have a repeat sigmoidoscopy performed at week 8. A food frequency questionnaire will be performed on week 0 and a food diary will be collected at week 2 and 12. A compliance questionnaire will be completed on weeks 2, 8and 12. A 24 hours recall will be collected at weeks 0, 2 and 6.

Patients in group 1 or 2 in remission from FT, may receive up to 2 rescue enemas during the 8 weeks of the study from their original donor.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Established diagnosis of UC, disease confined to the large intestine, involving the rectosigmoid for at least 3 months.
3. Age: 18 - 70 years ( inclusive)
4. Mild to Moderate active disease, SCCAI of ≥5 and <10 with endoscopic subscore≥2
5. Refractory to mesalamine 6 weeks, or steroids > 14 days, or immunomodulator 12 weeks or biologics at least 12 weeks therapy.
6. No use or stable use for 2 weeks of medical cannabis.

Inclusion criteria Comments:

1. Patients can enter the trial if they are on steroids if they have been treated for at least two weeks with 40 mg prednisone or an intravenous steroid such as methylprednisolone and still suffer from a mild to moderate active disease.

Exclusion Criteria:

1. Start of a new biologic in the previous 12 weeks.
2. Evidence for Clostridium difficile infection.
3. Any proven current infection such as CMV, positive stool culture or parasite.
4. Current Extra intestinal manifestation of UC such as active arthritis or primary sclerosing cholangitis (PSC).
5. Immune deficiency (other than drug induced).
6. Current use of a calcineurin inhibitor
7. Pregnancy.
8. Suspected toxic megacolon, guarding on palpation, or signs of peritoneal inflammation
9. Patients with other IBD unrelated disease such as autoimmune disorders, renal failure, fever or current infection (UTI, strep throat, pneumonia, etc), prior or current neoplasia
10. Fecal Transplantation in the last 6 months.
11. Fever >38
12. Participation in another clinical interventional trial
13. An active malignant disease or a prior malignancy during the previous 5 years (excluding skin BCC).
14. Inability or reluctance to use an enema.
15. Anticipation for antibiotic use within the study period (such as for elective surgery or dental treatment).
16. Acute severe UC in the past 3 months.
17. Presence of a pouch or pouchitis.
18. Patients > 60 years old using chronic medications except for the treatment for colitis.

Exclusion criteria Comments:

* Patients will be excluded from the analysis if during the study and after the initial fecal transplant they did not perform the enemas, used antibiotics prior to day 42. Patients who required additional therapy such as additional FMT, steroids biologics or immunomodulators during the first 8 weeks will be considered failures on an intention to treat basis.
* Patients with mayo< 2 at the baseline colonoscopy may receive the FMT and continue the follow up according to the protocol as an open lable based on the randomization. Those patients will be excluded from the final analysis.

Special populations (e.g children, unable to sign an informed consent, those under a guardian) and pregnant women will also be excluded.

Donors:

Donors will sign an informed consent and will be screened and included only if they satisfy the rigorous screening criteria of the protocol of the Ministry of Health of Israel for stool donors for Clostridium difficile infection which includes a list of medical and behavioral conditions as well as transmissible pathogens that need to be screened by history, anthropometry, blood and stool tests (available as supplement).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical remission | Day 56
  determined by Simple Clinical Colitis Activity Index (SCCAI) score <3 at week 8

SECONDARY OUTCOMES:
Improvement | Days 56 & 84
  Improvement in the Simple Clinical Colitis Activity Index (SCCAI) score at weeks 8 & 12 for each of the groups
Endoscopic resutls | Day 56
  Mayo endoscopic score <2 (for patients performing sigmoidoscopy)
Calprotectin | Day 56
  Calprotectin < 250 µg/g
The need for additional therapy or flare | Week 12
  According to the physician discretion
change in the microbiome compared to baseline. | For donor- day 14 and for recipient day 56
  According to analysis of fecal samples
endoscopic SCCAI | Day 56
  endoscopic SCCAI score at week 8 for each of the groups

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Principal Investigator — Wolfson Medical Center; Yona Avni, MD, Principal Investigator — Wolfson Medical Center
Locations (5):
- Saint-Antoine Hospital, Universite Pierre et Marie Curie, Paris, France
- Israel (2):
  - Wolfson Medical Center, Holon
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Humanitas Clinical and Research Center, Milan
  - Catholic University of the Secret Heart, Rome

REFERENCES:
- [Background] Sarbagili Shabat C, Scaldaferri F, Zittan E, Hirsch A, Mentella MC, Musca T, Cohen NA, Ron Y, Fliss Isakov N, Pfeffer J, Yaakov M, Fanali C, Turchini L, Masucci L, Quaranta G, Kolonimos N, Godneva A, Weinberger A, Kopylov U, Levine A, Maharshak N. Use of Faecal Transplantation with a Novel Diet for Mild to Moderate Active Ulcerative Colitis: The CRAFT UC Randomised Controlled Trial. J Crohns Colitis. 2022 Mar 14;16(3):369-378. doi: 10.1093/ecco-jcc/jjab165. PMID 34514495